CLINICAL TRIAL: NCT03860558
Title: Impact of Metabolic Health on Sperm Epigenetic Marks in Humans
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Joslin Diabetes Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2015-40
Record Dates: First submitted 2018-10-11; First posted 2019-03-04 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Overweight; Type 2 Diabetes Mellitus; Type 1 Diabetes Mellitus
MeSH Terms: conditions — Overweight; Diabetes Mellitus, Type 2; Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Lifestyle Intervention (Experimental): 20 overweight men with T1D or T2D will undergo an intensive 3 month lifestyle intervention program aimed at improving metabolic health, glycemic control, and body weight.
  Interventions: Other: Lifestyle Intervention
- No-Intervention Controls (Active Comparator): 10 overweight men with T1D or T2D will be assessed at baseline and at 3 months. They will not participate in a lifestyle intervention.
  Interventions: Other: No Intervention
- Healthy Controls (Active Comparator): 10 healthy men will be assessed at baseline and at 3 months. They will not participate in a lifestyle intervention.
  Interventions: Other: No Intervention

INTERVENTIONS:
Other: Lifestyle Intervention — Participants will undergo a 12-week multidisciplinary program for weight control and intensive diabetes management. The program includes adjustments to diabetes medications to enhance weight reduction and improve glycemia, dietary modification, and activity instructions.
  Arms: Lifestyle Intervention
Other: No Intervention — Participants will not undergo an intervention.
  Arms: Healthy Controls; No-Intervention Controls

SUMMARY:
This study is designed to evaluate whether epigenetic markers in overweight men with type 1 diabetes (T1D) or type 2 diabetes (T2D) can be improved with a 3 month lifestyle intervention or program focused in glycemic intervention.

DETAILED DESCRIPTION:
Parental history of diabetes confers substantial individual risk for development of obesity and diabetes. Obesity risk can be transmitted across generations, from parents or grandparents to children. Genomic variation explains only a portion of this risk. Epigenetic modulation through DNA methylation, histone modification, or by noncoding RNAs, provide mechanisms to regulate gene activity independent of DNA sequence by determining which genes are turned on or off in response to environment or disease. Epigenetic changes can be stable over the lifespan providing a mechanism through which environmental exposures may impart long-term effects on gene expression and phenotypic outcome.

The maternal intrauterine environment is now well recognized to modify obesity and T2D disease risk of offspring. Fetuses carried by women who are obese, have diabetes, or suffer from suboptimal nutrition are at increased risk of insulin resistance, obesity, T2D, and cardiovascular disease risk as adults. Studies in rodents also show that the health, metabolism, and prior environmental exposures of the male can also influence health of his offspring. Existing data provide powerful support for the hypothesis that current glucose levels and overall metabolic health of males can alter epigenetic marks in sperm and suggest a novel modifiable mechanism of transmission. However, much less is known about how human sperm epigenetic patterns change with nutritional and metabolic health, and whether these may ultimately impart differences in health of future generations. Thus, we are studying the impact of both type 1 and type 2 diabetes, and elevations in glucose common to both conditions, on human reproductive health and the sperm epigenome.

ELIGIBILITY:
Inclusion Criteria:

* Male, age 18-65 years
* Willing and able to provide informed consent and follow all study procedures, including providing sperm specimens 3 months apart.
* Type 1 or type 2 diabetes diagnosis confirmed by an endocrinologist (for participants in the diabetes groups)
* HbA1c > 7% (for participants in the diabetes groups)
* Overweight (BMI > 25 kg/m2) (for all groups, to ensure groups are similar)

Exclusion Criteria:

* Chronic kidney disease stage 4 or 5 (including end-stage renal disease);
* Hepatic disease, including serum alanine transaminase (ALT) or aspartate aminotransferase (AST) greater than or equal to 3 times the upper limit of normal; hepatic synthetic insufficiency as defined as serum albumin < 3.0 g/dL; or serum bilirubin > 2.0;
* Severe diabetic retinopathy;
* Congestive heart failure, New York Heart Association (NYHA) class II, III or IV;
* History of myocardial infarction, unstable angina or revascularization within the past 6 months;
* Active genitourinary infection;
* Testicular volume <12 mL (assessed using Prader orchidometer);
* Hypogonadism, defined as total testosterone <250 ng/dl;
* Hyperprolactinemia, defined as prolactin >18 ng/ml;
* Hyperestrogenism, defined as estradiol >42 pg/ml;
* Cryptorchidism;
* Cigarette smoking;
* Active alcohol abuse or substance abuse;
* Cancer (except localized non-melanoma skin cancers) or use of chemotherapy agents within 5 years;
* Use of nitrates or guanylate cyclase stimulators;
* Use of steroid hormones (including testosterone), other than inhalers for reactive airway disease

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2018-05-01 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Spermatozoa concentration | 1 year
  Sperm will be assessed for concentration, reported as total yield (millions per ml)

SECONDARY OUTCOMES:
Sperm DNA methylation, reported as genomic location of regions with methylation altered in response to intervention | 1 year
  We will utilize purified DNA (1.5 μg), sheared by sonication to obtain 200-700 bp fragments for subsequent library preparation for methylation-dependent immunoprecipitation and sequencing. Differentially methylated regions (DMR) are identified using methylated DNA immunoprecipitation coupled with next-generation sequencing (MEDIPS). DNA methylation is assessed using sliding windows (500 bp size, 200 bp shift). Regions with read ratios >1.5 or <0.67 and binomial p<0.0001 in independent biologically replicated comparisons are designated as DMR.
RNA Sequencing | 1 year
  RNA will be isolated from sperm samples and subjected to RNA sequencing to analyze the content of both of large messenger ribonucleic acid (mRNA)/noncoding RNA and small RNAs. Data will be analyzed to identify those species altered in response to intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- Joslin Diabetes Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sales VM, Ferguson-Smith AC, Patti ME. Epigenetic Mechanisms of Transmission of Metabolic Disease across Generations. Cell Metab. 2017 Mar 7;25(3):559-571. doi: 10.1016/j.cmet.2017.02.016. PMID 28273478
- [Derived] Su L, Dreyfuss JM, Ferraz Bannitz R, Wolfs D, Hansbury G, Richardson L, Charmant C, Patel J, Ginsburg ES, Racowsky C, Fore R, Efthymiou V, Desmond J, Goldfine A, Ferguson-Smith A, Pan H, Hivert MF, Isganaitis E, Patti ME. Type 2 diabetes impacts DNA methylation in human sperm. Clin Epigenetics. 2025 Mar 20;17(1):49. doi: 10.1186/s13148-025-01853-9. PMID 40108650